CLINICAL TRIAL: NCT02764541
Title: Palbociclib and Endocrine Therapy for LObular Breast Cancer Preoperative Study (PELOPS): A Randomized Phase II Study of Palbociclib With Letrozole Versus Letrozole Alone for Invasive Lobular Carcinoma and Invasive Ductal Carcinoma
Brief Title: Palbociclib and Endocrine Therapy for LObular Breast Cancer Preoperative Study (PELOPS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Otto Metzger, MD, Otto Metzger, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-052
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Results first posted 2023-08-31 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Invasive Lobular Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Lobular | interventions — Letrozole; Tamoxifen; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A Tamoxifen followed by Endocrine Therapy (Experimental): Tamoxifen is given in the Window of Treatment phase for 2 weeks followed by Endocrine Therapy for 24 weeks.
  Interventions: Drug: Tamoxifen; Drug: Endocrine Therapy
- Arm B Letrozole Followed By Endocrine Therapy (Experimental): Letrozole is given in the Window of Treatment phase for 2 weeks followed by Endocrine Therapy for 24 weeks.
  Interventions: Drug: Letrozole; Drug: Endocrine Therapy
- Tamoxifen Followed By Endocrine Therapy and Palbociclib (Experimental): Tamoxifen is given in the Window of Treatment phase for 2 weeks followed by Endocrine Therapy in combination with Palbociclib for 24 weeks.
  Interventions: Drug: Tamoxifen; Drug: Palbociclib; Drug: Endocrine Therapy
- Letrozole Followed By Endocrine Therapy and Palbociclib (Experimental): Letrozole is given in the Window of Treatment phase for 2 weeks followed by Endocrine Therapy in combination with Palbociclib for 24 weeks.
  Interventions: Drug: Letrozole; Drug: Palbociclib; Drug: Endocrine Therapy

INTERVENTIONS:
Drug: Letrozole
  Other Names: Femara
  Arms: Arm B Letrozole Followed By Endocrine Therapy; Letrozole Followed By Endocrine Therapy and Palbociclib
Drug: Tamoxifen
  Other Names: Soltanox
  Arms: Arm A Tamoxifen followed by Endocrine Therapy; Tamoxifen Followed By Endocrine Therapy and Palbociclib
Drug: Palbociclib
  Other Names: Ibrance
  Arms: Letrozole Followed By Endocrine Therapy and Palbociclib; Tamoxifen Followed By Endocrine Therapy and Palbociclib
Drug: Endocrine Therapy
  Other Names: Nolvadex

SUMMARY:
This research study is evaluating how well Breast Cancer responds to preoperative treatment with Endocrine treatment in combination with a drug called Palbociclib or Endocrine treatment alone as possible treatments for Hormone Receptor Positive Breast Cancer.

DETAILED DESCRIPTION:
This is an open label phase II neoadjuvant clinical trial of Palbociclib in combination with endocrine therapy for hormone receptor positive early-stage breast cancer. The planned sample size is 180 participants. The study includes a "window treatment" phase followed by a treatment phase. In the window phase, participants will be treated with a two-week course of tamoxifen (Arm A) or letrozole (Arm B). In the treatment phase participants will be randomized to receive endocrine therapy in combination with palbociclib (Arm C) or endocrine therapy alone (Arm D) for a total duration of 24 weeks. Premenopausal patients with either invasive lobular or ductal carcinoma will be eligible to enroll directly into the treatment phase of the study. The study has two co-primary objectives: 1) To evaluate the difference in anti-proliferative activity of letrozole versus tamoxifen measured by changes in Ki67 from baseline to research biopsy (day 15) within cohorts of hormone receptor positive breast cancer for patients with invasive lobular and ductal carcinoma. 2) To evaluate the pathologic complete response (pCR) of endocrine therapy plus palbociclib and of endocrine therapy alone in breast cancer patients diagnosed with hormone receptor positive invasive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Stage I to III histologically confirmed invasive carcinoma of the breast. A minimum tumor size of at least 1.5 cm determined by physical exam or imaging (whichever is larger) is required.
* Patients must have histologically confirmed hormone receptor positive (ER and/or PR), HER2 negative, invasive breast cancer. ER, PR and HER2 measurements should be performed according to institutional guidelines, in a CLIA-approved setting in the US or certified laboratories for Non-US regions. Cut-off values for positive/negative staining should be in accordance with current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines. Central confirmation is not required for ER, PR, or HER statuses.
* Patients with equivocal HER2 in situ hybridization results according to current ASCO/CAP guidelines are allowed, as long as the clinician has determined that they should be treated as HER2 negative.
* For the window phase: Patients must have histologically confirmed invasive lobular carcinoma or invasive ductal carcinoma. No central confirmation of histological subtype is necessary for enrollment.
* For the treatment phase: Patients with any histological subtype are eligible.
* Women 18 years of age. Men are not eligible.
* ECOG performance status 0 or 1
* Required laboratory values:

  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 10g/dL
  * Total serum bilirubin ≤ ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range in patients with documented Gilbert's Syndrome
  * Aspartate amino transferase (AST or SGOT) and alanine amino transferase (ALT or SGPT) ≤ 2.0 × institutional ULN
  * Serum creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with serum creatinine levels above institutional ULN
* Postmenopausal patients defined as no spontaneous menses ≥1 year (12 months) or post bilateral surgical oophorectomy. Premenopausal patients are eligible to participate provided they are considered in chemical menopause. Premenopausal patients should receive ongoing treatment with LHRH agonists (goserolin or leuprolide). Premenopausal patients must be enrolled directly into the treatment phase of the study.
* Patient must agree to the required research biopsies at baseline and after the two-week treatment with endocrine therapy in the initial part of the study ("window phase"); or at baseline and after two-week treated with endocrine therapy plus or minus palbociclib for those patients enrolled directly into the treatment phase of the study.
* Patients must be able and willing to swallow and retain oral medication without a condition that would interfere with enteric absorption.
* Breast imaging should include imaging of the ipsilateral axilla. For subjects with a clinically negative axilla, a sentinel lymph node biopsy will be performed either before or after preoperative therapy at the discretion of the subject's physicians. For subjects with a clinically positive axilla, a needle aspiration, core biopsy or SLN procedure will be performed to determine the presence of metastatic disease in the lymph nodes.
* Patients with multifocal or multicentric disease are eligible if the treating clinician has determined the patient should be treated as ER+ and HER2- negative.
* Bilateral breast cancers are allowed if the treating clinician has determined the patient should be treated as ER+ and HER2- negative.
* Serum or urine pregnancy test must be negative in women judged premenopausal within 7 days of randomization, or in women with amenorrhea of less than 12 months at time of randomization. Pregnancy testing does not need to be pursued in patients who are judged as postmenopausal before randomization, as determined by local practice, or who have undergone bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation.
* Premenopausal patients must agree to use adequate contraception for the duration of protocol treatment and for 6 months after the last treatment with palbociclib. Adequate contraception is defined as one highly effective form (i.e. abstinence, male or female sterilization) OR two effective forms (e.g. non-hormonal IUD and condom/occlusive cap with spermicidal foam / gel / film / cream/ suppository). Hormonal contraceptive methods are not allowed.
* Patients with a history of ipsilateral or contralateral DCIS are eligible.
* Patients may concurrently receive bisphosphonates or rank ligand inhibitors while on this study if necessary for treatment or prevention of osteopenia or osteoporosis. Prior treatment with LHRH agonists is allowed for premenopausal women. Topical vaginal estrogen therapy is allowable.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Concurrent therapy with other Investigational Products.
* Prior therapy with any CDK inhibitor.
* Patients with Stage IV breast cancer are not eligible. Baseline staging to document absence of metastatic disease is not required, however is recommended as determined by institutional practice (in patients where there may be a reasonable suspicion of advanced disease e.g., large tumors, clinically positive axillary lymph nodes, signs and symptoms). If performed, reports of these examinations must be available. Examination type for staging, i.e. X-ray, sonography, bone scans, CT, MRI, and/or PET-CT, is at the discretion of the investigator.
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to palbociclib.
* Patients receiving any medications or substances that are potent inhibitors or inducers of CYP3A isoenzymes within 7 days of randomization
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes, or psychiatric illness/social situations that would limit compliance with study requirements. Ability to comply with study requirements is to be assessed by each investigator at the time of screening for study participation.
* Pregnant women, or women of childbearing potential without a negative pregnancy test (serum or urine) within 7 days prior to randomization, irrespective of the method of contraception used, are excluded from this study because the effect of palbociclib on a developing fetus is unknown. Breastfeeding must be discontinued prior to study entry.
* Patients with a history of any malignancy are ineligible except for the following circumstances:

  * Patients with a malignancy history other than invasive breast cancer are eligible if they have no active malignancy and are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * Patients with the following cancers are eligible: ductal carcinoma in situ of the breast, cervical cancer in situ, and non-metastatic non-melanomatous skin cancers.
* Patients on combination antiretroviral therapy, i.e. those who are HIV-positive, are ineligible because of the potential for pharmacokinetic interactions or increased immunosuppression with palbociclib. HIV testing is not required, but patients must not be known to be HIV-positive.
* Patients receiving concurrent exogenous hormone therapy (hormone replacement therapy, oral or any other hormonal contraceptives such as hormonal contraceptive coil are not eligible.
* Patients are not eligible if they have previously received endocrine therapy within 5 years prior to diagnosis of the current malignancy. This includes use for prophylactic reasons, including treatment of osteoporosis or cancer prevention with tamoxifen, raloxifene, or AI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2031-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Otto Metzger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (11):
- United States (11):
  - Stamford Hospital, Stamford, Connecticut
  - Eastern Maine Medical Center, Brewer, Maine
  - Dana-Farber at St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - DF/BWCC at Milford Regional Medical Center, Milford, Massachusetts
  - DF/BWCC in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Lifespan, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss A, Jin Q, Tayob N, Wrabel E, DeMeo M, Carter J, Constantine M, Faggen M, Block C, Fenton MA, Lo KMS, Openshaw T, Yardley D, Kennedy L, Bedrosian I, Mittendorf EA, Jeselsohn R, Metzger Filho O, King TA. Axillary Management and Outcomes After Neoadjuvant Endocrine Therapy in the Randomized PELOPS Trial. Ann Surg Oncol. 2025 Nov 23. doi: 10.1245/s10434-025-18697-5. Online ahead of print. PMID 41276768
- [Derived] Weiss A, Revette A, Nava-Coulter B, Mittendorf EA, Filho OM, King TA. Surgeon Perspectives on Axillary Management Following Neoadjuvant Endocrine Therapy: Results from a Qualitative Substudy of the PELOPS Trial. Ann Surg Oncol. 2025 Nov 21. doi: 10.1245/s10434-025-18695-7. Online ahead of print. PMID 41272386
- [Derived] Hermida-Prado F, Xie Y, Sherman S, Nagy Z, Russo D, Akhshi T, Chu Z, Feit A, Campisi M, Chen M, Nardone A, Guarducci C, Lim K, Font-Tello A, Lee I, Garcia-Pedrero J, Canadas I, Agudo J, Huang Y, Sella T, Jin Q, Tayob N, Mittendorf EA, Tolaney SM, Qiu X, Long H, Symmans WF, Lin JR, Santagata S, Bedrosian I, Yardley DA, Mayer IA, Richardson ET, Oliveira G, Wu CJ, Schuster EF, Dowsett M, Welm AL, Barbie D, Metzger O, Jeselsohn R. Endocrine Therapy Synergizes with SMAC Mimetics to Potentiate Antigen Presentation and Tumor Regression in Hormone Receptor-Positive Breast Cancer. Cancer Res. 2023 Oct 2;83(19):3284-3304. doi: 10.1158/0008-5472.CAN-23-1711. PMID 37450351

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients withdrew consent before receiving intervention
Groups:
- Arm A Tamoxifen First, Then Arm C Endocrine With Palbociclib: Tamoxifen is given in the window phase for 2 weeks; Endocrine therapy in combination with Palbociclib are given in the treatment phase for 24 weeks
- Arm A Tamoxifen First, Then Arm D Endocrine Alone: Tamoxifen is given in the window phase for 2 weeks; Endocrine therapy alone is given in the treatment phase for 24 weeks
- Arm B Letrozole First, Then Arm C Endocrine With Palbociclib: Letrozole is given in the window phase for 2 weeks; Endocrine therapy in combination with Palbociclib are given in the treatment phase for 24 weeks
- Arm B Letrozole First, Then Arm D Endocrine Alone: Letrozole is given in the window phase for 2 weeks; Endocrine therapy alone is given in the treatment phase for 24 weeks
- Arm A Tamoxifen Only: Tamoxifen is given in the window phase for 2 weeks
- Arm B Letrozole Only: Letrozole is given in the window phase for 2 weeks
- Arm C Endocrine With Palbociclib Only: Endocrine therapy in combination with Palbociclib are given in the treatment phase for 24 weeks
- Arm D Endocrine Alone Only: Endocrine therapy alone is given in the treatment phase for 24 weeks
Period: Overall Study
Arm/Group | Arm A Tamoxifen First, Then Arm C Endocrine With Palbociclib | Arm A Tamoxifen First, Then Arm D Endocrine Alone | Arm B Letrozole First, Then Arm C Endocrine With Palbociclib | Arm B Letrozole First, Then Arm D Endocrine Alone | Arm A Tamoxifen Only | Arm B Letrozole Only | Arm C Endocrine With Palbociclib Only | Arm D Endocrine Alone Only
Started | 36 | 21 | 37 | 19 | 1 | 2 | 55 | 21
Completed | 33 | 20 | 36 | 16 | 0 | 0 | 52 | 18
Not Completed | 3 | 1 | 1 | 3 | 1 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Metastasis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Three Cycles completed before surgery | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Patient Compliance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Insurance reasons | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Tamoxifen First, Then Arm C Endocrine With Palbociclib | Arm A Tamoxifen First, Then Arm D Endocrine Alone | Arm B Letrozole First, Then Arm C Endocrine With Palbociclib | Arm B Letrozole First, Then Arm D Endocrine Alone | Arm A Tamoxifen Only | Arm B Letrozole Only | Arm C Endocrine With Palbociclib Only | Arm D Endocrine Alone Only | Total
Number analyzed (Participants) | 36 | 21 | 37 | 19 | 1 | 2 | 55 | 21 | 192
Age, Continuous [Median (Full Range); unit: years] | 64.0 [42.0 to 81.0] | 62.0 [53.0 to 80.0] | 64.0 [51.0 to 83.0] | 65.0 [50.0 to 77.0] | 56.0 [56.0 to 56.0] | 62.0 [58.0 to 66.0] | 49.0 [32.0 to 75.0] | 48.0 [33.0 to 56.0] | 57.0 [32.0 to 83.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 21 | 37 | 19 | 1 | 2 | 55 | 21 | 192
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 8
  Not Hispanic or Latino | 33 | 19 | 33 | 17 | 1 | 2 | 48 | 19 | 172
  Unknown or Not Reported | 3 | 1 | 3 | 1 | 0 | 0 | 4 | 0 | 12
Race [Count of Participants; unit: Participants]
  Black or African American | 5 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 11
  White | 31 | 20 | 33 | 18 | 1 | 2 | 47 | 17 | 169
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3
  More than one race | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 7
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Menopausal Status [Count of Participants; unit: Participants]
  Post-menopausal | 35 | 21 | 37 | 19 | 1 | 2 | 8 | 0 | 123
  Pre-menopausal | 1 | 0 | 0 | 0 | 0 | 0 | 47 | 21 | 69
Baseline Histology [Count of Participants; unit: Participants]
  Invasive Ductal | 14 | 11 | 19 | 10 | 0 | 0 | 29 | 9 | 92
  Invasive Lobular | 21 | 7 | 17 | 9 | 0 | 2 | 19 | 9 | 84
  Both | 1 | 3 | 1 | 0 | 1 | 0 | 7 | 2 | 15
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Baseline clinical N stage [Count of Participants; unit: Participants] — This is based on the diagnostic test and shows the extent the tumor spread to the lymph nodes. Higher stage is associated with worse outcome.
  Participants
    N0 | 19 | 11 | 19 | 10 | 1 | 2 | 28 | 12 | 102
    N1 | 17 | 9 | 17 | 8 | 0 | 0 | 21 | 9 | 81
    N2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
    N3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Unknown | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 5
Baseline clinical T stage [Count of Participants; unit: Participants] — This is based on the diagnostic test and describes the size and location of the tumor. Higher stage is associated with worse outcome.
  Participants
    T1a | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    T1b | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    T1c | 6 | 2 | 2 | 2 | 0 | 0 | 3 | 2 | 17
    T2 | 20 | 12 | 21 | 13 | 1 | 2 | 34 | 11 | 114
    T3 | 8 | 5 | 12 | 4 | 0 | 0 | 15 | 8 | 52
    T4 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 5
    Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Baseline Invasive Primary Breast Cancer Stage [Count of Participants; unit: Participants] — This stage was assigned by combining the tumor size/location, node, metastasis, tumor grade, and the results of ER/PR and HER2 testing results. Higher stage is associated with worse outcome.
  Participants
    I | 4 | 2 | 2 | 1 | 0 | 0 | 6 | 0 | 15
    II | 26 | 17 | 27 | 18 | 1 | 2 | 44 | 19 | 154
    III | 6 | 2 | 8 | 0 | 0 | 0 | 5 | 2 | 23
Surgery Type [Count of Participants; unit: Participants]
  Breast Conservation/Lumpectomy | 17 | 10 | 20 | 12 | 0 | 0 | 21 | 5 | 85
  Mastectomy | 17 | 10 | 17 | 5 | 0 | 0 | 31 | 13 | 93
  Missing | 2 | 1 | 0 | 2 | 1 | 2 | 3 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Difference in Anti-proliferative Activity of Patients Given Letrozole Versus Tamoxifen During the Window Phase
Description: Log fold change in anti-proliferative activity of Letrozole versus Tamoxifen within cohorts of hormone receptor positive breast cancer for patients with invasive lobular and ductal carcinoma during the window phase. Higher absolute value indicates larger change in the anti-proliferative activity
Time Frame: baseline to day 15
Population: Patients both not missing baseline and day15 Ki67 were included into the analysis population
Measure: Mean (Standard Deviation); unit: log fold-change
Groups:
- Tamoxifen With Invasive Ductal: Patients with invasive ductal/both histology receiving Tamoxifen in the window phase
- Letrozole With Invasive Ductal: Patients with invasive ductal/both histology receiving Letrozole in the window phase
- Tamoxifen With Invasive Lobular: Patients with invasive lobular histology receiving Tamoxifen in the window phase
- Letrozole With Invasive Lobular: Patients with invasive lobular histology receiving Letrozole in the window phase
Arm/Group | Tamoxifen With Invasive Ductal | Letrozole With Invasive Ductal | Tamoxifen With Invasive Lobular | Letrozole With Invasive Lobular
Number analyzed (Participants) | 27 | 28 | 25 | 25
log fold-change | -0.180 (2.5) | -1.304 (2.2) | -0.635 (2.5) | -1.944 (2.6)
Statistical Analysis 1: Comparison: Tamoxifen With Invasive Ductal vs Letrozole With Invasive Ductal; Test type: Equivalence — The hypothesis is that there is no difference in anti-proliferative activity of Letrozole vs Tamoxifen by measuring the fold-change in percent Ki67 from baseline to day15 in log scale within hormone receptor positive breast cancer patients with invasive ductal carcinoma; p = 0.0045, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tamoxifen With Invasive Lobular vs Letrozole With Invasive Lobular; Test type: Equivalence — The hypothesis is that there is no difference in anti-proliferative activity of Letrozole vs Tamoxifen by measuring the fold-change in percent Ki67 from baseline to day15 in log scale within hormone receptor positive breast cancer patients with invasive lobular carcinoma; p = 0.0161, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Pathologic Complete Response (pCR) of Patients Given Endocrine Therapy Plus Palbociclib and of Endocrine Therapy Alone During the Treatment Phase
Description: Residual Cancer Burden index (RCB) between hormone receptor positive invasive breast cancer patients given endocrine therapy plus palbociclib (Arm C) and endocrine therapy alone (Arm D). RCB score is used to assess the response to neoadjuvant chemotherapy in breast cancer patients and is in a scale of 0 to infinity. Higher RCB score indicates more tumor burden remaining, thus worse outcome.
Time Frame: day 15 to 24 weeks
Population: Patients with treatment and surgery are included into the analysis population
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Arm C Endocrine With Palbociclib: Endocrine therapy in combination with Palbociclib are given in the treatment phase for 24 weeks.
- Arm D Endocrine Therapy Alone: Endocrine therapy alone is given in the treatment phase for 24 weeks
Arm/Group | Arm C Endocrine With Palbociclib | Arm D Endocrine Therapy Alone
Number analyzed (Participants) | 128 | 60
score on a scale | 2.88 [0.00 to 4.83] | 2.88 [0.03 to 4.71]
Statistical Analysis 1: Comparison: Arm C Endocrine With Palbociclib vs Arm D Endocrine Therapy Alone; Test type: Equivalence — The hypothesis is that there is no difference of pathologic response measured by RCB index between Arm C and Arm D; p = 0.9288, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Odds Ratio of Achieving Cell Cycle Arrest at the End of Window Phase
Description: Odds Ratio of Achieving Cell Cycle Arrest at the end of Window Phase in hormone receptor positive invasive breast cancer patients given Tamoxifen vs Letrozole. Cell cycle arrest is defined to be percentage of Ki67<2.7
Time Frame: baseline to day 15
Population: Patients both not missing baseline and day15 Ki67 were included into the analysis population
Measure: Number (95% Confidence Interval); unit: odds ratio
Groups:
- Tamoxifen vs Letrozole in Invasive Ductal Patients: Patients with invasive ductal/both histology receiving Tamoxifen vs Letrozole in the window phase
- Tamoxifen vs Letrozole in Invasive Lobular Patients: Patients with invasive lobular histology receiving Tamoxifen vs Letrozole in the window phase
Arm/Group | Tamoxifen vs Letrozole in Invasive Ductal Patients | Tamoxifen vs Letrozole in Invasive Lobular Patients
Number analyzed (Participants) | 55 | 50
odds ratio | 0.26 [0.08 to 0.89] | 0.60 [0.19 to 1.9]

4. Secondary Outcome: Change in RCB Index Between Arm C and Arm D During the Treatment Phase
Description: The estimate of RCB index change for patients who receive both endocrine and Palbociclib instead of endocrine alone, but have the same lymph node status, tumor size and menopausal status. RCB score is used to assess the response to neoadjuvant chemotherapy in breast cancer patients and is in a scale of 0 to infinity. Higher RCB score indicates more tumor burden remaining, thus worse outcome.
Time Frame: day 15 to 24 weeks
Population: Patients with treatment and surgery are included into the analysis population
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Endocrine With Palbociclib: Endocrine therapy in combination with Palbociclib
- Endocrine Alone: Endocrine therapy alone
Arm/Group | Endocrine With Palbociclib | Endocrine Alone
Number analyzed (Participants) | 128 | 60
units on a scale | 2.88 [0.00 to 4.83] | 2.88 [0.03 to 4.71]
Statistical Analysis 1: Comparison: Endocrine With Palbociclib vs Endocrine Alone; Test type: Equivalence — The hypothesis is that there is no difference of pathologic response measured by RCB index between Arm C and Arm D; p = 0.920, Regression, Linear; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.29 to 0.32]

5. Secondary Outcome: Number of Participants With RCB Response in Arm C and Arm D During the Treatment Phase
Description: RCB response is defined as RCB-0 or RCB-I; RCB not response is defined as RCB-II or RCB-III Residual Cancer Burden (RCB) considers residual disease in the tumor bed and lymph nodes after NAC, generating a continuous score which is then grouped into four categories: RCB-0, RCB-I, RCB-II and RCB-III. Higher RCB group reflects more tumor burden remaining, thus worse outcome
Time Frame: day 15 to 24 weeks
Population: Patients with treatment and surgery are included into the analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm C Endocrine With Palbociclib | Arm D Endocrine Therapy Alone
Number analyzed (Participants) | 128 | 60
Participants | 10 | 3
Statistical Analysis 1: Comparison: Arm C Endocrine With Palbociclib vs Arm D Endocrine Therapy Alone; Test type: Equivalence — The hypothesis is that there is no difference of RCB response rate between Arm C and Arm D; p = 0.758, Fisher Exact

6. Secondary Outcome: Percentage of Participants With Clinical Response in Arm C and Arm D in the Treatment Phase
Description: Percentage of Participants with Clinical Response in Arm C and Arm D in Breast cancer patients diagnosed with hormone receptor positive invasive breast cancer; Clinical response rate is defined as the number of partial and complete responses after preoperative endocrine therapy plus palbociclib (Arm C) and of endocrine therapy alone (Arm D)
Time Frame: day 15 to 24 weeks
Population: Patients with treatment and surgery are included into the analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Arm C Endocrine With Palbociclib | Arm D Endocrine Therapy Alone
Number analyzed (Participants) | 128 | 60
percentage of participants | 57.8 | 43.3

ADVERSE EVENTS:
Time Frame: The adverse event data were collected after starting the first dose of study treatment and before 30 days following the last administration of study treatment or study discontinuation/termination (up to 27 weeks), whichever is earlier.
Description: Serious AEs are defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. AEs were collected without specifying which phase they occurred in and are reported by patients' treatment sequence, which is consistent with the participant flow and considered as the most feasible way.
Arm/Group | Arm A Tamoxifen First, Then Arm C Endocrine With Palbociclib | Arm A Tamoxifen First, Then Arm D Endocrine Alone | Arm B Letrozole First, Then Arm C Endocrine With Palbociclib | Arm B Letrozole First, Then Arm D Endocrine Alone | Arm A Tamoxifen Only | Arm B Letrozole Only | Arm C Endocrine With Palbociclib Only | Arm D Endocrine Alone Only
All-Cause Mortality (participants affected / at risk) | 1/36 | 2/21 | 0/37 | 1/19 | 0/1 | 0/2 | 3/55 | 1/21
Serious Adverse Events (participants affected / at risk) | 3/36 | 3/21 | 14/37 | 0/19 | 0/1 | 0/2 | 21/55 | 0/21
Other Adverse Events (participants affected / at risk) | 36/36 | 21/21 | 37/37 | 18/19 | 0/1 | 1/2 | 55/55 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A Tamoxifen First, Then Arm C Endocrine With Palbociclib (N=36) | Arm A Tamoxifen First, Then Arm D Endocrine Alone (N=21) | Arm B Letrozole First, Then Arm C Endocrine With Palbociclib (N=37) | Arm B Letrozole First, Then Arm D Endocrine Alone (N=19) | Arm A Tamoxifen Only (N=1) | Arm B Letrozole Only (N=2) | Arm C Endocrine With Palbociclib Only (N=55) | Arm D Endocrine Alone Only (N=21)
Neutrophil count decreased (Investigations) | 3 | 0 | 13 | 0 | 0 | 0 | 18 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A Tamoxifen First, Then Arm C Endocrine With Palbociclib (N=36) | Arm A Tamoxifen First, Then Arm D Endocrine Alone (N=21) | Arm B Letrozole First, Then Arm C Endocrine With Palbociclib (N=37) | Arm B Letrozole First, Then Arm D Endocrine Alone (N=19) | Arm A Tamoxifen Only (N=1) | Arm B Letrozole Only (N=2) | Arm C Endocrine With Palbociclib Only (N=55) | Arm D Endocrine Alone Only (N=21)
Anemia (Blood and lymphatic system disorders) | 6 | 0 | 4 | 0 | 0 | 0 | 6 | 0
Hypothyroidism (Endocrine disorders) | 5 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Blurred vision (Eye disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 2 | 5 | 1 | 0 | 0 | 9 | 4
Diarrhea (Gastrointestinal disorders) | 8 | 4 | 7 | 1 | 0 | 0 | 15 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9 | 2 | 7 | 6 | 0 | 0 | 4 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 10 | 0 | 10 | 1 | 0 | 0 | 15 | 0
Nausea (Gastrointestinal disorders) | 13 | 5 | 7 | 3 | 0 | 0 | 14 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 27 | 9 | 26 | 10 | 0 | 1 | 34 | 6
Fever (General disorders) | 4 | 0 | 0 | 1 | 0 | 0 | 3 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 7 | 3 | 9 | 6 | 0 | 0 | 8 | 0
Pain (General disorders) | 5 | 4 | 3 | 4 | 0 | 0 | 6 | 5
Breast infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 4 | 1 | 0 | 0 | 4 | 0
Skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 4 | 0 | 3 | 1 | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 3 | 0 | 0 | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 3 | 0 | 0 | 0 | 3 | 0
Cholesterol high (Investigations) | 2 | 2 | 3 | 5 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 28 | 0 | 23 | 0 | 0 | 0 | 43 | 0
Platelet count decreased (Investigations) | 5 | 0 | 4 | 0 | 0 | 0 | 9 | 0
White blood cell decreased (Investigations) | 5 | 0 | 3 | 0 | 0 | 0 | 12 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9 | 11 | 6 | 0 | 0 | 10 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 4 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 0 | 0 | 0 | 7 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 3 | 0 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 6 | 0 | 0 | 0 | 5 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 4 | 0 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 5 | 3 | 4 | 0 | 0 | 0 | 11 | 0
Headache (Nervous system disorders) | 8 | 5 | 6 | 3 | 0 | 0 | 20 | 4
Anxiety (Psychiatric disorders) | 8 | 5 | 6 | 2 | 0 | 0 | 17 | 4
Depression (Psychiatric disorders) | 5 | 4 | 5 | 4 | 0 | 0 | 8 | 3
Insomnia (Psychiatric disorders) | 8 | 5 | 12 | 7 | 0 | 0 | 18 | 8
Breast pain (Reproductive system and breast disorders) | 8 | 7 | 5 | 3 | 0 | 0 | 5 | 3
Vaginal dryness (Reproductive system and breast disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 5 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 2 | 0 | 0 | 5 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 6 | 2 | 1 | 0 | 0 | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 1 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 21 | 17 | 14 | 10 | 0 | 0 | 37 | 17
Hypertension (Vascular disorders) | 15 | 6 | 13 | 8 | 0 | 0 | 13 | 5
Bloating (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 3 | 0
Edema limbs (General disorders) | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7 | 1 | 0 | 0 | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 5 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 2 | 0 | 0 | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0 | 0 | 0 | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 3 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 3 | 0
Body odor (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 3
Blood prolactin abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT02764541/Prot_SAP_001.pdf